CLINICAL TRIAL: NCT03072849
Title: Early Detection and Management of Bronchiolitis Obliterans Syndrome Following Pediatric Hematopoietic Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Jennifer Schneiderman, MD, MD, MS, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: SCT 1214 BOS
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Bronchiolitis Obliterans Syndrome
Keywords: Pediatrics; Airflow obstruction; Chronic graft-vs-host disease; Bronchiolitis obliterans syndrome
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Respiratory Physiological Phenomena; Fluticasone; Inhalation; Azithromycin; montelukast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Stem Cell Transplant Recipients: Pediatric patients ages 6-18 years who have received allogenic hematopoietic stem cell transplant for any reason.
  Interventions: Procedure: Pulmonary function testing; Drug: FAM Therapy

INTERVENTIONS:
Procedure: Pulmonary function testing — Each enrolled patient will receive pulmonary function testing every three months. Pulmonary function testing includes spirometry, plethysmography, and diffusion capacity measurements.
  Other Names: PFT; Spirometry; Plethysmography; Diffusion capacity
Drug: FAM Therapy — All patients who have evidence of early airflow obstruction on pulmonary function testing will be started on FAM therapy. Early airflow obstruction is defined by a FEV1 decline of ≥10% predicted in addition to a FVC <0.8.
  Other Names: Fluticasone (Inhaled); Azithromycin; Montelukast

SUMMARY:
This study aims to determine whether or not early spirometric detection and management of obstructive lung disease with combined fluticasone/azithromycin/montelukast therapy (FAM) can attenuate declining lung function, prevent the development of bronchiolitis obliterans, and improve patient outcomes following hematopoietic stem cell transplant.

DETAILED DESCRIPTION:
Bronchiolitis obliterans syndrome (BOS) is an inflammatory condition of the lungs that leads to obstructive physiology, irreversible fibrosis of terminal bronchioles, and obliteration of the small airways. In both children and adults, the prevalence of BOS is approximately 6% in those with chronic graft-vs-host disease (cGVHD), although this may be a gross underestimation given current diagnostic guidelines. Once diagnosed, the prognosis is extremely unfavorable. BOS carries a mortality rate of approximately 40-60%, with a five year survival rate of 13%.

Early on, BOS is symptomatically silent. Once symptoms are present, there is a high likelihood of irreversible disease regardless of the combination of immune suppression used. Given these circumstances, early diagnosis is of utmost importance, and can be characterized by an isolated and subclinical decline in lung function. Recent studies have suggested that early decline in lung function on pulmonary function testing (PFT) may be representative of developing BOS.

Due to the lack of consistent screening and diagnostic criteria, many patients with evolving BOS elude a timely diagnosis, thereby jeopardizing their chance of survival. In response, several experts have recommended frequent PFT screening and a modified, less stringent set of diagnostic criteria with the goal of establishing earlier diagnosis and timely intervention.

Traditionally, treatment of BOS has included aggressive immunosuppression, leaving patients at risk for life-threatening invasive infections, multi-system co-morbidities, and the threat of lung transplantation. Recent studies have demonstrated that early management with agents such as inhaled corticosteroids (ICS), macrolides, and leukotriene receptor antagonists (LTRA) can lead to improvements in both lung function and clinical symptoms.

This study aims to evaluate the utility of frequent and routine pulmonary surveillance in pediatric patients who have undergone allogenic HSCT. Our prospective study design provides a novel framework for the implementation of standardized lung function screening every three months in the first two years following HSCT. With this, we hypothesize that standardized PFT screening will improve diagnostic sensitivity and allow for earlier intervention in patients with evolving airway obstruction and BO.

This study also aims to evaluate the efficacy of inhaled fluticasone, azithromycin, and montelukast (FAM therapy) in the management of early airflow obstruction in pediatric patients following allogenic HSCT. Early airflow obstruction is defined by pulmonary function testing (FEV1 decline of ≥10% predicted with a FVC <0.8). With this, we hypothesize that FAM therapy will attenuate the progression of airflow obstruction and improve lung function in those with irreversible airflow obstruction at one and two years when compared to historical controls.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: Patients undergoing myeloablative allogenic hematopoietic stem cell transplant for any indication (both malignant and non-malignant) are eligible.
2. Graft: Eligible patients will have one or more of the following donor stem cell sources:

   * Bone marrow
   * Placental blood (umbilical cord blood)
   * Cytokine mobilized peripheral blood
3. Eligible patients will have one of the following sources of donor stem cells:

   * HLA matched family member
   * Partially matched family member (mismatched for a single HLA locus at A, B, C or DR)
   * Fully HLA matched or partially mismatched unrelated marrow or peripheral blood stem cells (per institutional donor selection standards)
   * HLA matched or partially mismatched (at least 4/6 match at A, B, DR) cord blood.
4. Conditioning Regimen: Patients expecting to receive any type of myeloablative HSCT conditioning regimen are eligible.
5. Prior therapies: Patients undergoing stem cell transplant of any kind.
6. Required laboratory parameters: Patients able to adequately perform pulmonary function testing per ATS/ERS guidelines, as determined by the enrolling investigator and trained respiratory therapists.
7. The patient and/or the patient's legally authorized guardian must acknowledge in writing that consent to become a study subject has been obtained in accordance with the institutional policies approved by the U.S. Department of Health and Human Services. Informed consent must be signed prior to registration on study.

Exclusion Criteria:

1. Subjects with a previous solid organ transplant.
2. Recurrent or progressive malignancy requiring anti-cancer therapy.
3. Subjects with evidence of underlying obstructive pulmonary disease prior to transplant (clinical history of asthma or baseline FEV1 <80% predicted with FEV1/FVC <80%).
4. Known history of allergy or intolerance to Montelukast, Zafirleukast, Azithromycin, Erythromycin, Clarithromycin, Prednisone, or Sirolimus.
5. Chronic supplemental oxygen requirement or hypoxemia <92% SpO2.
6. Clinical asthma (variable and recurrent symptoms of airflow obstruction and airway hyper-responsiveness).
7. Pregnancy or nursing: All females of childbearing age must have a negative serum or urine pregnancy test <7 days before study drug administration.
8. Chronic treatment with any inhaled steroid for >1 month in past three months.
9. Treatment with montelukast or zafirukast for >1 month in past three months.
10. Treatment with systemic steroids for >1 month in past three months.
11. Treatment with any FDA non-approved study medication within the past four weeks. Off label treatment with FDA approved medication is allowed.
12. Evidence of any viral, bacterial, or fungal infection involving the lung and not responding to appropriate treatment.
13. Inability to perform pulmonary function testing (PFT), as determined by the enrolling investigator or PFT lab.
14. Any condition that, in the opinion of the enrolling investigator, would interfere with the subject's ability to comply with the study requirements.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients undergoing allogenic hematopoietic stem cell transplant
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2015-04; Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Lung function | 2 years
  Change in lung function at 12 and 24 months post-HSCT
Survival | 2-4 years
  Overall survival at 2 years post-HSCT

SECONDARY OUTCOMES:
Risk factor assessment | 2 years
  To identify risk factors for the development of BOS

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chien JW, Martin PJ, Gooley TA, Flowers ME, Heckbert SR, Nichols WG, Clark JG. Airflow obstruction after myeloablative allogeneic hematopoietic stem cell transplantation. Am J Respir Crit Care Med. 2003 Jul 15;168(2):208-14. doi: 10.1164/rccm.200212-1468OC. Epub 2003 Mar 20. PMID 12649126
- [Background] Bergeron A, Belle A, Chevret S, Ribaud P, Devergie A, Esperou H, Ades L, Gluckman E, Socie G, Tazi A. Combined inhaled steroids and bronchodilatators in obstructive airway disease after allogeneic stem cell transplantation. Bone Marrow Transplant. 2007 May;39(9):547-53. doi: 10.1038/sj.bmt.1705637. Epub 2007 Mar 12. PMID 17351647
- [Background] Bashoura L, Gupta S, Jain A, Couriel DR, Komanduri KV, Eapen GA, Safdar A, Broglio KR, Adachi R, Dickey BF. Inhaled corticosteroids stabilize constrictive bronchiolitis after hematopoietic stem cell transplantation. Bone Marrow Transplant. 2008 Jan;41(1):63-7. doi: 10.1038/sj.bmt.1705877. Epub 2007 Oct 15. PMID 17934530
- [Background] Kaya Z, Weiner DJ, Yilmaz D, Rowan J, Goyal RK. Lung function, pulmonary complications, and mortality after allogeneic blood and marrow transplantation in children. Biol Blood Marrow Transplant. 2009 Jul;15(7):817-26. doi: 10.1016/j.bbmt.2009.03.019. PMID 19539213
- [Background] Norman BC, Jacobsohn DA, Williams KM, Au BK, Au MA, Lee SJ, Moravec CK, Chien JW. Fluticasone, azithromycin and montelukast therapy in reducing corticosteroid exposure in bronchiolitis obliterans syndrome after allogeneic hematopoietic SCT: a case series of eight patients. Bone Marrow Transplant. 2011 Oct;46(10):1369-73. doi: 10.1038/bmt.2010.311. Epub 2010 Dec 6. PMID 21132024
- [Background] Hildebrandt GC, Fazekas T, Lawitschka A, Bertz H, Greinix H, Halter J, Pavletic SZ, Holler E, Wolff D. Diagnosis and treatment of pulmonary chronic GVHD: report from the consensus conference on clinical practice in chronic GVHD. Bone Marrow Transplant. 2011 Oct;46(10):1283-95. doi: 10.1038/bmt.2011.35. Epub 2011 Mar 28. PMID 21441964
- [Background] Pulsipher MA, Skinner R, McDonald GB, Hingorani S, Armenian SH, Cooke KR, Gracia C, Petryk A, Bhatia S, Bunin N, Nieder ML, Dvorak CC, Sung L, Sanders JE, Kurtzberg J, Baker KS. National Cancer Institute, National Heart, Lung and Blood Institute/Pediatric Blood and Marrow Transplantation Consortium First International Consensus Conference on late effects after pediatric hematopoietic cell transplantation: the need for pediatric-specific long-term follow-up guidelines. Biol Blood Marrow Transplant. 2012 Mar;18(3):334-47. doi: 10.1016/j.bbmt.2012.01.003. Epub 2012 Jan 14. PMID 22248713
- [Background] Majhail NS, Rizzo JD, Lee SJ, Aljurf M, Atsuta Y, Bonfim C, Burns LJ, Chaudhri N, Davies S, Okamoto S, Seber A, Socie G, Szer J, Van Lint MT, Wingard JR, Tichelli A; Center for International Blood and Marrow Transplant Research; American Society for Blood and Marrow Transplantation; European Group for Blood and Marrow Transplantation; Asia-Pacific Blood and Marrow Transplantation Group; Bone Marrow Transplant Society of Australia and New Zealand; East Mediterranean Blood and Marrow Transplantation Group; Sociedade Brasileira de Transplante de Medula Ossea. Recommended screening and preventive practices for long-term survivors after hematopoietic cell transplantation. Bone Marrow Transplant. 2012 Mar;47(3):337-41. doi: 10.1038/bmt.2012.5. PMID 22395764
- [Background] Gassas A, Craig-Barnes H, Dell S, Doyle J, Schechter T, Sung L, Egeler M, Palaniyar N. Chest health surveillance utility in the early detection of bronchiolitis obliterans syndrome in children after allo-SCT. Bone Marrow Transplant. 2013 Jun;48(6):814-8. doi: 10.1038/bmt.2012.228. Epub 2012 Nov 19. PMID 23165500
- [Background] Prais D, Sinik MM, Stein J, Mei-Zahav M, Mussaffi H, Steuer G, Hananya S, Krauss A, Yaniv I, Blau H. Effectiveness of long-term routine pulmonary function surveillance following pediatric hematopoietic stem cell transplantation. Pediatr Pulmonol. 2014 Nov;49(11):1124-32. doi: 10.1002/ppul.22944. Epub 2013 Nov 4. PMID 24574432
- [Background] Madanat-Harjuoja LM, Valjento S, Vettenranta K, Kajosaari M, Dyba T, Taskinen M. Pulmonary function following allogeneic stem cell transplantation in childhood: a retrospective cohort study of 51 patients. Pediatr Transplant. 2014 Sep;18(6):617-24. doi: 10.1111/petr.12313. Epub 2014 Jul 7. PMID 25041660